CLINICAL TRIAL: NCT00848549
Title: A Randomized, Double-Blind Extension Study To Assess The Long-Term Safety And To Explore The Long-Term Efficacy Of Zonisamide As Monotherapy In Newly Diagnosed Partial Seizures
Brief Title: Assessing The Long-Term Safety And To Explore The Long-Term Efficacy Of Zonisamide As Monotherapy In Newly Diagnosed Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2090-E044-314; 2008-001159-23 (EudraCT Number)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; Monotherapy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ZNS (Active Comparator)
  Interventions: Drug: Zonisamide
- CBZ (Active Comparator)
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Zonisamide — Subjects will start on the same dose that was achieved at the end of study E2090-E044-310. Maximum daily dose allowable is 500 mg; the minimum daily dose allowable is 200 mg. During the study, subjects will be titrated up or down depending on seizure-free status or intolerability/adverse events, respectively. Should a dose outside of the maximum be required the subject will be with drawn and gradually down titrated by 100 mg per week.
  Other Names: Zonegran
  Arms: ZNS
Drug: Carbamazepine — Subjects will start on the same dose that was achieved at the end of study E2090-E044-310. Maximum daily dose allowable is 1200 mg; the minimum daily dose allowable is 400 mg. During the study, subjects will be titrated up or down depending on seizure-free status or intolerability/adverse events respectively. Should a dose outside of the maximum be required the subject will be with drawn and gradually down titrated by 200 mg per week.
  Arms: CBZ

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability and to explore the long-term efficacy of zonisamide as monotherapy treatment in subjects with newly diagnosed partial seizures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed study E2090-E044-310.
2. Subject is able and willing to give written informed consent.
3. Female subjects without childbearing potential (two years post-menopausal, bilateral oophorectomy or tubal ligation, complete hysterectomy) are eligible. Female subjects of childbearing potential must be non-pregnant, non-lactating and abide by one of the following medically acceptable contraceptive measures: oral contraceptive pill, contraceptive injections, implants or patches, intrauterine device in place for at least three months, vasectomised partner or abstinence throughout the study and for one month after discontinuation of study medication. When the contraceptive pill is used, this should contain no less than 50 μg oestrogen.
4. The subject is able and willing to follow the investigational study procedures, maintain a seizure diary and report adverse events.

Exclusion Criteria:

1. Subject has a history of a significant or currently uncontrolled disease that will contraindicate the use of the study drugs or interfere with the conduct of this study and/or the assessment of safety and efficacy of the study drugs.
2. Subject has a body weight <40 kg.
3. Subject has a newly occurring progressive malignancy during study E2090-E044-310 (excluding a history of non-metastasized and adequately treated cutaneous squamous cell carcinoma).
4. Subject has developed a psychiatric illness or mood disorder requiring electro-convulsive or drug therapy within the previous 6 months and is considered uncontrolled; history of suicide attempt, alcohol or drug abuse, chronic treatment with benzodiazepines or barbiturates.
5. Subject is currently taking carbonic anhydrase inhibitors.
6. Subject developed pancreatitis, nephrolithiasis or hypercalcuria, clinically significant laboratory abnormalities, stroke or uncontrolled hypertension during study E2090-E044-310.
7. Subject is currently taking monoamine oxidase inhibitors (MAOIs) or any other excluded medications (see protocol section 9.9.3).
8. Subject has a history of allergy to carbamazepine or to zonisamide or to any of their ingredients or to sulphonamides.
9. Subject has developed a bone marrow depression, low platelet count or other blood dyscrasias.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Baulac, Principal Investigator — Hopital de la Pitie-Saltpetriere
Locations (110):
- Australia (8):
  - Camperdown, New South Wales
  - Bedford Park, South Australia
  - Clayton, Victoria
  - Fitzroy, Victoria
  - Heidelberg West, Victoria
  - Parkville, Victoria
  - Perth, Western Australia
  - Queensland
- Aalborg, Denmark
- France (4):
  - Béthune
  - Dijon
  - Paris
  - Saint-Etienne
- Germany (6):
  - Berlin
  - Bochum
  - Düsseldorf
  - Munich
  - Schwerin
  - Westerstede
- Greece (3):
  - Athens
  - Pátrai
  - Thessaloniki
- Hungary (6):
  - Budapest
  - Debrecen
  - Gyula
  - Hódmezővásárhely
  - Nyregyhaza
  - Zalaegerszeg-Poozva
- India (7):
  - Bangalore
  - Hyderabad
  - Koturpuram, Chennai
  - Madurai, Tamil Nadu
  - Mumbai
  - New Delhi
  - Pune
- Italy (10):
  - Catanzaro
  - Messina
  - Milan
  - Monza (MI)
  - Orbassano
  - Pavia
  - Rome
  - Siena
  - Turin
  - Udine
- Podgorica, Montenegro
- Poland (9):
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Sosnowiec
  - Szczecin
  - Warsaw
- Russia (6):
  - Kaliningrad
  - Kazan'
  - Madrid
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Serbia (7):
  - Belgrade
  - Kragujevac
  - Kruševac
  - Niš
  - Novi Sad
  - Sombor
  - Subotica
- Slovakia (7):
  - Bratislava
  - Brezno
  - Košice
  - NoveZamky
  - Spitalska 6
  - Vranov nad Topľou
  - Žilina
- South Africa (8):
  - Bellair
  - Berea
  - Parktown
  - Pretoria
  - Richards Bay
  - Sandton
  - Tygerberg
  - Umhlanga
- South Korea (3):
  - Anyang
  - Seoul
  - Wŏnju
- Spain (8):
  - Alicante
  - Barcelona
  - Cruces (Vizcaya)
  - Madrid
  - Málaga
  - Oviedo
  - Seville
  - Zaragoza
- Sweden (3):
  - Gothenburg
  - Linköping
  - Lund
- Switzerland (3):
  - Basel
  - Bern
  - Sankt Gallen
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Taoyuan District
  - Yongkang District
- United Kingdom (6):
  - Bristol
  - Cardiff
  - Glasgow
  - Liverpool
  - Tooting
  - Treliske

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E2090-E044-314 is a double-blind extension of E2090-E044-310 (NCT00477295) "base study." Assessment of eligibility took place at the Study Entry Visit (SEV), which was the same day as their final visit of Study 310. Subjects remained on the same investigational product as they were randomized to in Study 310 until unblinding of that study.
Groups:
- Zonisamide: Subjects received the same study drug to which they had been randomized in the core study phase and remained on their final dose for the start of the extension phase (between 200 mg and 500 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
- Carbamazepine: Subjects received the same study drug to which they had been randomized in the core study phase and remained on their final dose for the start of the extension phase (between 400 mg and 1200 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
Period: E2090-E044-310 (Base Study) Disposition
Arm/Group | Zonisamide | Carbamazepine
Started | 282 | 301
Completed | 161 | 192
Not Completed | 121 | 109
Not completed — Adverse Event | 31 | 35
Not completed — Withdrawal by Subject | 35 | 24
Not completed — Lack of Efficacy | 23 | 23
Not completed — Protocol Violation | 3 | 8
Not completed — Physician Decision | 4 | 5
Not completed — Lost to Follow-up | 21 | 11
Not completed — Other | 4 | 3
Period: E2090-E044-310 (Base Study) Transition
Arm/Group | Zonisamide | Carbamazepine
Started | 161 | 192
Completed | 137 | 158
Not Completed | 24 | 34
Not completed — Chose not to enter 314 Extension study | 24 | 34
Period: E2090-E044-314 (Extension Study)
Arm/Group | Zonisamide | Carbamazepine
Started | 137 | 158
Completed | 120 | 134
Not Completed | 17 | 24
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Other | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Carbamazepine | Total
Number analyzed (Participants) | 282 | 301 | 583
Age, Continuous [Mean (Standard Deviation); unit: years]
  Base Study 310 (NCT00477295, n=583) | 37.1 (16.33) | 35.6 (15.50) | 36.35 (15.92)
  Extension Study 314 (NCT00848549, n=295) | 37.8 (16.13) | 34.4 (14.93) | 36.1 (15.53)
Sex/Gender, Customized [Number; unit: participants]
  Female (Base Study 310, NCT00477295) | 107 | 128 | 235
  Male (Base Study 310, NCT00477295) | 174 | 172 | 346
  Female (Extension Study 314, NCT00848549) | 57 | 59 | 116
  Male (Extension Study 314, NCT00848549) | 80 | 99 | 179

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Remaining in the Study at Each Visit
Description: The retention rate is defined as the percentage of subjects remaining on the study at each visit, starting from the first dose of study drug in the extension phase.
Time Frame: At 3, 6, 9, 12, 15, 18, 21, 24, and 27 months
Population: The Intent-to-Treat (ITT) Population is defined as all subjects who received at least one dose of investigational product(IP)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Zonisamide: Subjects received the same study drug to which they had been randomized in the base study phase and remained on their final dose for the start of the extension phase (between 200 mg and 500 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
- Carbamazepine: Subjects received the same study drug to which they had been randomized in the base study phase and remained on their final dose for the start of the extension phase (between 400 mg and 1200 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 137 | 158
Percentage of Participants
  3 months | 95.6 [92.2 to 99.1] | 93.7 [89.8 to 97.5]
  6 months | 87.6 [82.0 to 93.2] | 84.2 [78.4 to 89.9]
  9 months | 76.6 [69.5 to 83.8] | 75.3 [68.5 to 82.1]
  12 months | 58.4 [50.1 to 66.7] | 61.4 [53.7 to 69.0]
  15 months | 38.7 [30.5 to 46.9] | 43.7 [35.9 to 51.5]
  18 months | 27.7 [20.2 to 35.3] | 27.8 [20.8 to 34.9]
  21 months | 13.1 [7.4 to 18.8] | 12.7 [7.4 to 17.9]
  24 months | 5.8 [1.9 to 9.8] | 2.5 [0.1 to 5.0]
  27 months | 1.5 [0.0 to 3.5] | 0.6 [0.0 to 1.9]

2. Secondary Outcome: Time to Drop-out Due to Lack of Efficacy
Description: Lack of efficacy was if the subject had poor seizure control (defined as experiencing a seizure despite being on the maximum dose for = 2 weeks). The subject could withdraw at any time due to lack of efficacy.
Time Frame: Week 1 to Week 109 (in core study) and Month 1 to Month 27 (in extension study)
Population: 310 ITT Population (combined ITT Population from basecore study and extension phase). 24 participants were discontinued in each arm due to lack of efficacy; these were the participants that were evaluated in this outcome.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 24 | 24
Days | 297.9 (170.03) | 289.0 (108.93)

3. Secondary Outcome: Time to Drop-out Due to Adverse Event (AE)
Description: Adverse events in study subjects included any change in the subject's condition.
  This includes symptoms, physical findings, or clinical syndromes. All AEs that occurred after signing of informed consent through the last visit and for 15 days following study drug discontinuation were captured on the AE Case Report Form (CRF).
Time Frame: Week 1 to Week 109 (in base study) and Month 1 to Month 27 (in extension study)
Population: 310 ITT Population (33 participants were discontinued in the Zonisamide arm and 35 were discontinued in the Carbamazepine arm; these were the participants evaluated for this outcome)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 33 | 35
Days | 131.9 (166.90) | 97.2 (114.47)

4. Secondary Outcome: Percentage of Participants That Are Seizure Free for at Least 24 Month Consecutive Period in the Base Study and Extension Phase
Description: The number of participants that have remained seizure free for at least a 24 month consecutive period from the start of the Flexible Dosing Period (FDP: the period following the Titration Period and leading into the Maintenance Period) in the base study through the treatment period of this study. Seizure freedom was defined as the absence of all seizure regardless of seizure type.
Time Frame: Week 5 to Week 109 (in base study) and Month 1 to Month 27 (in extension phase)
Population: 310 ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 281 | 300
Percentage of Participants | 32.3 [26.5 to 38.0] | 35.2 [29.5 to 40.9]

5. Secondary Outcome: Change From Baseline in Quality of Life Assessed by Quality of Life in Epilepsy-Problems Questionnaire (QOLIE-31-P) Overall Score at Each Visit
Description: The QOLIE-31-P is a 31-item questionnaire evaluating a participant's QOL perception in 7 domains: seizure worry,emotional well being,energy/fatigue, cognitive functioning, medication effects, social functioning,overall QOL. The overall score is derived by weighing and then summing the 7 domain scores. Precoded numeric values for some domains are such that a higher number reflects a more favorable health state; others are such that a higher number reflects a less favorable state. Precoded values are converted to 0-100 point scores; higher converted scores always reflect better QOL.
Time Frame: Weeks 0, 26, 52, 78 and 117
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Zonisamide | Carbamazepine
Number analyzed (Participants) | 137 | 158
Score on a scale
  Week 0 | 4.697 (16.254) | 7.101 (13.781)
  Week 26 | 6.101 (16.566) | 10.956 (14.940)
  Week 52 | 8.602 (14.326) | 11.687 (13.653)
  Week 78 | 4.287 (15.566) | 1.902 (13.495)
  Week 117 | -0.292 (17.332) | 15.849 (12.302)

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent form through the Final Visit/Early Termination Visit and for 15 days following study drug discontinuation.
Description: Adverse events were assessed at clinical visits based on the subject's diary, vitals, weight, physical examination, neurological exam, and laboratory evaluations.
Groups:
- Zonisamide (Extension Study 314, NCT00848549): Subjects received the same study drug to which they had been randomized in the core study phase and remained on their final dose for the start of the extension phase (between 200 mg and 500 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
- Carbamazepine (Extension Study 314, NCT00848549): Subjects received the same study drug to which they had been randomized in the core study phase and remained on their final dose for the start of the extension phase (between 400 mg and 1200 mg per day). Flexible dosing was permitted as symptoms changed as long as it stayed within the dosing range.
- Zonisamide (Base Study 310, NCT00477295): The starting dose in this arm was zonisamide 100mg daily. The dose during the Titration Period (4 weeks) ranged from 100 to 200mg daily. During the Flexible Dosing Period (FDP), the subjects were given doses ranging from 300 to 500mg daily or if they could not tolerate that dose, were allowed one down-titration or were withdrawn. If the subjects remained seizure-free for 26 weeks by the end of FDP (the subject was allowed 3 chances to achieve this), they entered the Maintenance Period (26 weeks), where they remained on the same dose they were taking at the end of the FDP.
- Carbamazepine (Base Study 310, NCT00477295): The starting dose in this arm was carbamazepine 200mg daily. The dose during the Titration Period (4 weeks) ranged from 200 to 400mg daily. During the Flexible Dosing Period (FDP), the subjects were given doses ranging from 600 to 1200mg daily or if they could not tolerate that dose, were allowed one down-titration or were withdrawn. If the subjects remained seizure-free for 26 weeks by the end of FDP (the subject was allowed 3 chances to achieve this), they entered the Maintenance Period (26 weeks), where they remained on the same dose they were taking at the end of the FDP.
Arm/Group | Zonisamide (Extension Study 314, NCT00848549) | Carbamazepine (Extension Study 314, NCT00848549) | Zonisamide (Base Study 310, NCT00477295) | Carbamazepine (Base Study 310, NCT00477295)
Serious Adverse Events (participants affected / at risk) | 7/137 | 7/158 | 15/281 | 17/300
Other Adverse Events (participants affected / at risk) | 12/137 | 10/158 | 72/281 | 69/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (Extension Study 314, NCT00848549) (N=137) | Carbamazepine (Extension Study 314, NCT00848549) (N=158) | Zonisamide (Base Study 310, NCT00477295) (N=281) | Carbamazepine (Base Study 310, NCT00477295) (N=300)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Unwanted pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Partial seizures with secondary generalization (Nervous system disorders) | 0 | 0 | 0 | 4
Complex partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Typhoid fever (Infections and infestations) | 0 | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (Extension Study 314, NCT00848549) (N=137) | Carbamazepine (Extension Study 314, NCT00848549) (N=158) | Zonisamide (Base Study 310, NCT00477295) (N=281) | Carbamazepine (Base Study 310, NCT00477295) (N=300)
Weight Decreased (Investigations) | 8 | 0 | 19 | 0
Headache (Nervous system disorders) | 6 | 10 | 29 | 37
Somnolence (Nervous system disorders) | 0 | 0 | 17 | 23
Dizziness (Nervous system disorders) | 0 | 0 | 11 | 23
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 22 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No